CLINICAL TRIAL: NCT04228458
Title: Does Thermal Imaging Correlate With Musculoskeletal Examination in the Identification of Inflamed Joints in Children and Young People With Juvenile Idiopathic Arthritis? A Prospective Diagnostic Accuracy Study
Brief Title: ThermRheum Version 1
Acronym: ThermRheum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH-13-067d
Record Dates: First submitted 2020-01-08; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal Imaging (Experimental): Thermal Imaging acquisition
  Interventions: Device: Thermal Imaging

INTERVENTIONS:
Device: Thermal Imaging — Testing the effectiveness of using a Thermal Imaging camera in participants with Juvenile Arthritis.

SUMMARY:
Childhood arthritis is a diagnosis made by clinicians based upon their clinical examination, during which patients are assessed for signs of swelling, warmth and restricted movement of the joints using the sensation of touch. Clinicians use investigations such as blood tests and scans which may be costly, associated with waiting times, can cause the patient stress or anxiety. Patients with childhood arthritis can often present with flares of their condition even when on medical treatment, which may require further investigations to determine the nature of the problem. Studies in adult Rheumatology have demonstrated that a thermal imaging camera (which detects heat given off by the body) can be useful in assessing for signs of inflammation in arthritis. The use of this camera could provide an alternative to the tests described; it does not require any contact with the patient, is quick and easy to use, and does not emit any radiation. The investigators hope that this pilot study will demonstrate that thermal imaging can be used to complement the standardised assessments of joint inflammation as done routinely in clinic and may lead to further work comparing thermal imaging with other tests such as MRI scanning and ultra-sound.

The investigators will recruit 20-50 children with arthritis affecting either knee or ankle joints. The investigators will use a highly sensitive thermal imaging camera to take pictures and short video recordings of each ankle and knee joint, recording skin temperature and colour. The investigators will compare this with the clinicians' assessment of whether the knee and ankle joints are inflamed or not. The investigators are interested in finding out whether the information recorded using the camera mirrors the assessment made by the clinician.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of:

* Poly-articular JIA
* Oligo-articular JIA
* Psoriatic JIA
* Enthesitis-related JIA

Exclusion Criteria:

CYP below 4 years of age (pGALS is validated for school-age children and patients will be required to remain still during TI process)

Ongoing active/chronic infection requiring hospitalisation or treatment with intravenous antibiotics within 30 days of recruitment, or oral antibiotics within 14 days of recruitment

History of active tuberculosis of less than 6 months treatment or untreated latent tuberculosis

Soft tissue infection, injury or fracture of the affected joint which could confound the TI signature

Presence of any inflammatory skin condition (including, but not limited to Eczema and Psoriasis) which may be in close proximity to or overlying the joint

Presence of any other diagnosis which could cause arthritis including systemic-JIA (associated systemic inflammation may affect skin temperature independently of arthritis) or undifferentiated-JIA (excluded to ensure homogeneity of the sample investigated)

Non-English speaking patients and/or parent(s)/guardian(s)

Non-consenting CYP, or parent(s)/guardian(s)

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Correlation between Thermal Imaging and changes in skin temperature | 30 minutes
  Correlation between Thermal Imaging and changes in skin temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Childrens NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No